CLINICAL TRIAL: NCT02287324
Title: Immediate Effects of Cervical Spine Manipulation on Gait Parameters in Individuals With and Without Mechanical Neck Pain
Brief Title: Effects of Cervical Spine Manipulation on Gait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Emilio J Puentedura, PT, DPT, PhD, Principal Investigator, University of Nevada, Las Vegas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: UNLV-1303-4418
Record Dates: First submitted 2014-03-04; First posted 2014-11-10 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Cervicalgia
Keywords: Cervicalgia
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manipulation (Active Comparator): High velocity low amplitude thrust joint manipulation to the cervical spine
  Interventions: Procedure: Manipulation
- Manual Contact (Placebo Comparator): Manual contact to suboccipital region of the cervical spine for 5 minutes
  Interventions: Procedure: Manual Contact

INTERVENTIONS:
Procedure: Manipulation
  Arms: Manipulation
Procedure: Manual Contact
  Arms: Manual Contact

SUMMARY:
The purpose of the study is to see if manipulation of the neck will change the way people who may or may not have neck pain, walk under differing conditions.

DETAILED DESCRIPTION:
Volunteers in this study will be asked to do the following: 1) complete a series of questionnaires about health status and undergo physical screening of neck to make sure that manipulation will not be harmful; 2) walk in socks or bare feet across a computerized mat under 3 conditions - normal walking pace, walking while looking up and down repeatedly; and walking while looking left and right repeatedly; 3) have one of 2 manual therapy interventions to the neck; 4) repeat the walking across the computerized mat under those same 3 conditions.

The 2 randomly assigned interventions are: cervical manipulation, or cervical contact. If assigned the manipulation, volunteers will lie face up and the trained therapist will move the joints in the neck in a gentle, but short and sharp manner which may produce a slight 'pop' or 'click'. If volunteers are assigned the cervical contact, they will lie on their back and the trained therapist will gently hold the head and neck for 45 to 60 seconds as they quietly relax.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers may or may not have mechanical neck pain
2. Aged 18 to 70 years
3. If neck pain is present, must have Neck Disability Index score of at least 10 out of 50 points

Exclusion Criteria:

1. 'Red flag' items indicated in Neck Medical Screening Questionnaire such as history of a tumor, bone fracture, metabolic diseases, Rheumatoid Arthritis, osteoporosis, severe atherosclerosis, prolonged history of steroid use, etc.
2. History of neck whiplash injury
3. Diagnosis from physician of cervical spinal stenosis (narrowing of spinal canal) or presence of symptoms (pain, pins and needles, numbness) down both arms
4. Presence of central nervous system involvement such as exaggerated reflexes, changes in sensation in the hands, muscle wasting in the hands, impaired sensation of the face, altered taste, and presence of abnormal reflexes
5. Evidence of neurological signs consistent with nerve root entrapment (pinched nerve in the neck)
6. Prior surgery to neck or upper back
7. A medical condition which may influence assessment of pain or pressure pain thresholds (i.e. taking analgesics, sedatives, history of substance abuse, or cognitive deficiency)
8. Diagnosis from your physician of fibromyalgia syndrome
9. Currently pregnant, or could be pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Gait Parameters - Composite Score | Up to 10 minutes after intervention
  A composite score derived from specific gait parameters which include stride length, step length, step width, cadence

SECONDARY OUTCOMES:
Global Rating of Change Scale | Up to 10 minutes after intervention
  Global rating of perceived change

CONTACTS AND LOCATIONS:
Locations (1):
- UNLV, Las Vegas, Nevada, United States